CLINICAL TRIAL: NCT01131728
Title: A Randomized, Open Label, Two Treatment, Two Period, Two Sequence, Single Dose, Crossover, Bioequivalence Study of Naproxen Sodium 220 mg + Pseudoephedrine HCL 120 mg ER Tablets and Aleve Cold and Sinus® Under Fasting Conditions.
Brief Title: Bioequivalence Study of Naproxen Sodium 220 mg & Pseudoephedrine HCl 120 mg ER Tablets of Dr. Reddy's Under Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: M.S. Mohan / Vice President, R&D, Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 391/04
Record Dates: First submitted 2010-05-26; First posted 2010-05-27 (Estimated); Last update posted 2010-06-14 (Estimated); Status verified 2010-06

CONDITIONS: Healthy
Keywords: Bioequivalence; Crossover; Naproxen Sodium and Pseudoephedrine Hydrochloride
MeSH Terms: interventions — Naproxen; Pseudoephedrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Naproxen Sodium & Pseudoephedrine HCl (Experimental): Naproxen Sodium 220 mg and Pseudoephedrine Hydrochloride 120 mg ER Tablets of Dr. Reddy's Laboratories.
  Interventions: Drug: Naproxen Sodium & Pseudoephedrine HCl
- Aleve Cold and Sinus (Active Comparator): Aleve Cold and Sinus(Naproxen Sodium 220 mg and Pseudoephedrine Hydrochloride 120 mg Extended Release Tablets).
  Interventions: Drug: Naproxen Sodium & Pseudoephedrine HCl

INTERVENTIONS:
Drug: Naproxen Sodium & Pseudoephedrine HCl — Naproxen Sodium 220 mg and Pseudoephedrine Hydrochloride 120 mg Extended Release Tablets
  Other Names: Aleve Cold and Sinus

SUMMARY:
The purpose of this study is to assess the bioequivalence of Naproxen sodium 220 mg + Pseudoephedrine Hydrochloride 120 mg Extended Release tablets of with Aleve Cold and Sinus in healthy adult human subjects, under fasting conditions.

DETAILED DESCRIPTION:
Open randomized, two treatment, two period, two sequence, single dose, crossover study of 26 healthy human adult subjects under fasting conditions with a washout period of 14 days.

ELIGIBILITY:
Inclusion Criteria:

Subjects must fulfill all of the following criteria to be considered for inclusion into this study:

* Subjects will provide written informed consent.
* Subjects must be healthy human beings within 18-45 years of age (inclusive) weighing at least 50 kg.
* Subjects must be within ±15% of ideal body weight in relation to height according to Life Insurance Corporation of India height-weight chart for non- medical cases.
* Subjects must be of normal health as determined by medical history and physical examination performed within 21 days prior to the commencement of the study.
* Have normal ECG, X-ray and vital signs.
* Availability of subject for the entire study period and willingness to adhere to protocol requirements as evidenced by written informed consent.

If subject is a female volunteer and

* Is of child bearing potential practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), such as condoms, foams, jellies. diaphragm,intrauterine device (IUD), or abstinence.
* Is postmenopausal for at least 1 year.
* Is surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy has been performed on the subject.

Exclusion Criteria:

The subjects will be excluded under following conditions:

History or presence of significant:

* Cardiovascular, pulmonary, hepatic, renal, hematological, gastrointestinal, endocrine,immunologic, dermatologic, musculoskeletal, neurological or psychiatric disease.
* Alcohol dependence, alcohol abuse or drug abuse within past one year.
* Moderate to heavy smoking (>10 cigarettes/day) or consumption of tobacco products.
* Asthma, urticaria or other allergic type reactions after taking any medication.

Subjects who through completion of the study, would have donated in excess of

* 500 ml of blood in 14 days, or
* 500 - 800ml of blood in 14 days (unless approved by the Principal Investigator)
* 1000 ml of blood in 90 days
* 1250 ml of blood in 120 days
* 1500 ml of blood in 180 days
* 2000 ml of blood in 270 days
* 2500 ml of blood in 1 year Subjects who have participated in another clinical trial within 3 months of study start.

Subjects who have:

* Systolic blood pressure less than 90 mm of Hg and higher than 150 mm of Hg
* Diastolic blood pressure less than 60 mm of Hg and more than 95 mm of Hg. Minor deviations (1-3 mm Hg) at check-in may be acceptable at the discretion of the physician/investigator.
* Pulse rate below 50/min. and above 105/min. Female volunteers demonstrating a positive pregnancy screen or currently breast-feeding.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2004-07; Primary Completion 2004-08 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Bioequivalence based on Cmax and AUC parameters | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Sandhya Ravi, MBBS, MS., Principal Investigator — Lotus Labs Pvt. Ltd.,
Locations (1):
- Lotus Labs Private Limited, Bangalore, Karnataka, India